CLINICAL TRIAL: NCT00930059
Title: A PHASE 2 MULTICENTER, DOUBLE BLIND, PLACEBO CONTROLLED, PARALLEL GROUP STUDY OF PF-04447943 IN SUBJECTS WITH MILD TO MODERATE ALZHEIMER'S DISEASE
Brief Title: A Study Of PF-04447943 Compared To Placebo In Subjects With Mild To Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B0401005; 2009-012179-82 (EudraCT Number)
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; PF-04447943; efficacy; safety; plasma concentrations
MeSH Terms: conditions — Alzheimer Disease | interventions — 6-(4-methyl-1-(pyrimidin-2-ylmethyl)pyrrolidin-3-yl)-1-(tetrahydro-2H-pyran-4-yl)-1,5-dihydro-4H-pyrazolo(3,4-d)pyrimidin-4-one

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PF-04447943 (Experimental)
  Interventions: Drug: PF-04447943
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04447943 — tablets, 25 mg every 12 hours for 12 wks
  Arms: PF-04447943
Drug: Placebo — matching placebo tablets, every 12 hours for 12 wks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of PF-04447943 compared to placebo on cognitive, behavioral and overall symptoms of Alzheimer's disease; evaluate the safety and tolerability of PF-0444793 compared to placebo; and determine the levels of PF-04447943 in the plasma over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate Alzheimer's disease (MMSE 14-26)
* Good general health (such controlled conditions as Type 2 diabetes and hypertension allowed)

Exclusion Criteria:

* Use of acetylcholinesterase inhibitors (donepezil, rivastigmine, or galantamine) or memantine within 12 weeks of the start of the study
* Significant cardiovascular disease in the past 6 months
* Illness other than Alzheimer's disease that could contribute to cognitive impairment
* History of stroke or seizure disorder

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2009-09-10 (Actual); Primary Completion 2010-09-22 (Actual); Study Completion 2010-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (44):
- United States (22):
  - Neurology Clinic, PC, Northport, Alabama
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Southwestern Research Incorporated, Glendale, California
  - Pacific Coast Imaging (for Imaging only), Newport Beach, California
  - The Southwest Institute for Clinical Research, Inc., Rancho Mirage, California
  - Pacific Research Network (Satellite Site), San Diego, California
  - Pacific Research Network, Inc. (Satellite Site), Vista, California
  - MD Clinical, Hallandale, Florida
  - Compass Research, LLC, Orlando, Florida
  - Berma Research Group, Plantation, Florida
  - Joliet Center for Clinical Research, Joliet, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Agewell, Indianapolis, Indiana
  - Four Rivers Clinical Research, Inc., Paducah, Kentucky
  - Advanced MRI, Lake Charles, Louisiana
  - Lake Charles Clinical Trials, LLC, Lake Charles, Louisiana
  - Neurocare, Inc., Newton, Massachusetts
  - Neurobehavioral Research Inc, Cedarhurst, New York
  - Behavioral Medical Research of Staten Island, Staten Island, New York
  - University of Pittsburgh Alzheimer's Disease Research Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Alzheimer's Disease and Memory Disorders Center, Providence, Rhode Island
  - Neurology Clinic, PC, Cordova, Tennessee
- Canada (5):
  - Medical Arts Health Research Group, Kelowna, British Columbia
  - Hamilton Health Sciences, Hamilton, Ontario
  - Kawartha Regional Memory Clinic, Peterborough, Ontario
  - Neuro Rive Sud Clinic, Greenfield Park, Quebec
  - Diex Recherche Inc., Sherbrooke, Quebec
- Chile (8):
  - Psicomed Estudios Clinicos, Antofagasta, Antofagasta
  - Hospital Base Valdivia, Valdivia, Los Ríos Region
  - Centro Doctora Lissette Duque, Providencia, RM
  - Psicomedica Research Group, Santiago, RM
  - Hospital Del Salvador, Santiago, RM
  - Neuroconsult, Santiago, RM
  - Especialidades Medicas L y S, Santiago, RM
  - Neuropsicologia Ltda., La Florida, Santiago Metropolitan
- Czechia (9):
  - Fakultni nemocnice, Hradec Králové
  - Pardubicka krajska nemocnice, a.s., Pardubice
  - Pragtis, s.r.o., Prague
  - Fakultni nemocnice v Motole, Prague
  - Psychiatry Trial, s.r.o., Prague
  - Psychiatricka ambulance, Prague
  - Neurologie - EEG, s.r.o, Prague
  - Centrum neurologicke pece, s.r.o., Rychnov nad Kněžnou
  - Psychiatricka ambulance, Strakonice

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0401005&StudyName=A%20Study%20Of%20PF-04447943%20Compared%20To%20Placebo%20In%20Subjects%20With%20Mild%20To%20Moderate%20Alzheimer%27s%20Disease

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matched to PF-04447943 tablet orally twice daily for 12 weeks.
- PF-04447943: PF-04447943 25 milligram (mg) tablet orally twice daily for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | PF-04447943
Started | 100 | 91
Completed | 92 | 79
Not Completed | 8 | 12
Not completed — Death | 1 | 0
Not completed — Did not meet entrance criteria | 1 | 1
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Other | 1 | 0
Not completed — 1 site terminated by sponsor | 1 | 1
Not completed — Adverse Event | 1 | 6

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who consumed at least 1 dose of randomized study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-04447943 | Total
Number analyzed (Participants) | 100 | 91 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.5 (7.5) | 73.6 (8.2) | 73.5 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 58 | 122
  Male | 36 | 33 | 69

OUTCOME MEASURES:

1. Primary Outcome: Alzheimer's Disease Assessment Scale-Cognitive Subscale 70 (ADAS-Cog 70) Score at Baseline
Description: ADAS-cog is a structured scale assessing the severity of cognitive impairment in Alzheimer's disease. It comprises of following 11 items (range): word recall (0-10), naming objects and fingers (0-5), following commands (0-5), constructional praxis (0-5), ideational praxis (0-5), orientation (0-8), word recognition (0-12), recall of test instructions (0-5), spoken language ability (0-5), word-finding difficulty (0-5), comprehension of spoken language (0-5). Total ADAS-cog 70 score was sum of all items and ranged from 0 (least impairment) to 70 (most severe impairment), higher score indicating worse cognition.
Time Frame: Baseline (Day 1)
Population: FAS included all participants who consumed at least 1 dose of randomized study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-04447943
Number analyzed (Participants) | 100 | 91
units on a scale | 21.87 (10.42) | 22.66 (10.39)

2. Primary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale 70 (ADAS-Cog 70) at Week 12
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: FAS included all participants who consumed at least 1 dose of randomized study medication. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | PF-04447943
Number analyzed (Participants) | 93 | 80
units on a scale | -1.60 (0.50) | -1.91 (0.54)
Statistical Analysis 1: Comparison: Placebo vs PF-04447943; Least squares (LS) mean difference and p-values were based on analysis of covariance (ANCOVA) on change from baseline with treatment, baseline value, scheduled visit and visit by treatment interaction as covariates, and participant effect as random effect; Test type: Superiority; p = 0.3353, ANCOVA — The primary test of significance was 1-sided, and a nominal Type I error rate a = 0.05 was employed; LS mean difference = -0.31, 90% CI 2-sided [-1.52 to 0.90], Standard Error of Mean 0.73

3. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale 70 (ADAS-Cog 70) at Week 3, 6 and 9
Description: as for outcome 1
Time Frame: Baseline, Week 3, 6, 9
Population: FAS included all participants who consumed at least 1 dose of randomized study medication. "Number analyzed" signifies those participants who were evaluable for this measure at the specified time points for each arm, respectively.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | PF-04447943
Number analyzed (Participants) | 100 | 91
units on a scale
  Change at Week 3: number analyzed (Participants) | 100 | 89
  Change at Week 3 | -1.36 (0.49) | -1.16 (0.52)
  Change at Week 6: number analyzed (Participants) | 96 | 83
  Change at Week 6 | -1.17 (0.50) | -1.53 (0.53)
  Change at Week 9: number analyzed (Participants) | 97 | 82
  Change at Week 9 | -2.05 (0.50) | -2.68 (0.53)
Statistical Analysis 1: Comparison: Placebo vs PF-04447943; Change at Week 3: LS mean difference and p-values were based on ANCOVA on change from baseline with treatment, baseline value, scheduled visit and visit by treatment interaction as covariates, and participant effect as random effect; Test type: Superiority; p = 0.6073, ANCOVA — No adjustments made for multiple comparisons; LS mean difference = 0.20, 90% CI 2-sided [-0.99 to 1.38], Standard Error of Mean 0.72
Statistical Analysis 2: Comparison: Placebo vs PF-04447943; Change at Week 6: LS mean difference and p-values were based on ANCOVA on change from baseline with treatment, baseline value, scheduled visit and visit by treatment interaction as covariates, and participant effect as random effect; Test type: Superiority; p = 0.3086, ANCOVA — No adjustments made for multiple comparisons; LS mean difference = -0.36, 90% CI 2-sided [-1.56 to 0.84], Standard Error of Mean 0.73
Statistical Analysis 3: Comparison: Placebo vs PF-04447943; Change at Week 9: LS mean difference and p-values were based on ANCOVA on change from baseline with treatment, baseline value, scheduled visit and visit by treatment interaction as covariates, and participant effect as random effect; Test type: Superiority; p = 0.1970, ANCOVA — No adjustments made for multiple comparisons; LS mean difference = -0.62, 90% CI 2-sided [-1.82 to 0.58], Standard Error of Mean 0.73

4. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I)
Description: CGI-I is a 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale.
Time Frame: Week 3, 6, 9, 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | PF-04447943
Number analyzed (Participants) | 100 | 91
units on a scale
  Week 3: number analyzed (Participants) | 100 | 89
  Week 3 | 3.64 (0.10) | 3.70 (0.10)
  Week 6: number analyzed (Participants) | 96 | 84
  Week 6 | 3.51 (0.10) | 3.58 (0.11)
  Week 9: number analyzed (Participants) | 97 | 82
  Week 9 | 3.63 (0.10) | 3.45 (0.11)
  Week 12: number analyzed (Participants) | 93 | 80
  Week 12 | 3.53 (0.10) | 3.32 (0.11)
Statistical Analysis 1: Comparison: Placebo vs PF-04447943; Week 3: Inferential statistics were based on linear model with fixed effects for visit (nominal scale) and visit by treatment interaction, and a random effect for participant; Test type: Superiority; p = 0.6547, Linear model — No adjustments made for multiple comparisons; LS mean difference = 0.06, 90% CI 2-sided [-0.18 to 0.29], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Placebo vs PF-04447943; Week 6: Inferential statistics were based on linear model with fixed effects for visit (nominal scale) and visit by treatment interaction, and a random effect for participant; Test type: Superiority; p = 0.7020, Linear model — No adjustments made for multiple comparisons; LS mean difference = 0.08, 90% CI 2-sided [-0.16 to 0.31], Standard Error of Mean 0.14
Statistical Analysis 3: Comparison: Placebo vs PF-04447943; Week 9: Inferential statistics were based on linear model with fixed effects for visit (nominal scale) and visit by treatment interaction, and a random effect for participant; Test type: Superiority; p = 0.1138, Linear model — No adjustments made for multiple comparisons; LS mean difference = -0.17, 90% CI 2-sided [-0.41 to 0.06], Standard Error of Mean 0.14
Statistical Analysis 4: Comparison: Placebo vs PF-04447943; Week 12: Inferential statistics were based on linear model with fixed effects for visit (nominal scale) and visit by treatment interaction, and a random effect for participant; Test type: Superiority; p = 0.0816, Linear model — No adjustments made for multiple comparisons; LS mean difference = -0.20, 90% CI 2-sided [-0.44 to 0.04], Standard Error of Mean 0.15

5. Secondary Outcome: Neuropsychiatric Inventory (NPI) Total Score at Baseline
Description: NPI total score evaluates disturbances in 12 behavioral domains: delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, motor disturbance, appetite/eating and night time behavior. NPI total score ranged from 0 (minimum severity) to 144 (maximum severity); higher score indicates greater behavioral disturbances.
Time Frame: Baseline
Population: FAS included all participants who consumed at least 1 dose of randomized study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-04447943
Number analyzed (Participants) | 100 | 91
units on a scale | 12.16 (12.86) | 10.67 (11.28)

6. Secondary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Total Score at Week 3, 6, 9 and 12
Description: as for outcome 5
Time Frame: Baseline, Week 3, 6, 9, 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | PF-04447943
Number analyzed (Participants) | 100 | 91
units on a scale
  Change at Week 3: number analyzed (Participants) | 100 | 89
  Change at Week 3 | -2.02 (0.66) | -1.33 (0.70)
  Change at Week 6: number analyzed (Participants) | 97 | 84
  Change at Week 6 | -2.61 (0.66) | -1.76 (0.71)
  Change at Week 9: number analyzed (Participants) | 97 | 82
  Change at Week 9 | -3.44 (0.66) | -2.49 (0.72)
  Change at Week 12: number analyzed (Participants) | 93 | 80
  Change at Week 12 | -2.70 (0.67) | -2.86 (0.72)
Statistical Analysis 1: Comparison: Placebo vs PF-04447943; Change at Week 3: LS mean difference and p-value were based on ANCOVA on change from baseline with treatment, baseline value, scheduled visit and visit by treatment interaction as covariates, and participant effect as random effect; Test type: Superiority; p = 0.7634, ANCOVA — No adjustments have been made for multiple comparisons; LS mean difference = 0.69, 90% CI 2-sided [-0.89 to 2.27], Standard Error of Mean 0.96
Statistical Analysis 2: Comparison: Placebo vs PF-04447943; Change at Week 6: LS mean difference and p-value were based on ANCOVA on change from baseline with treatment, baseline value, scheduled visit and visit by treatment interaction as covariates, and participant effect as random effect; Test type: Superiority; p = 0.8077, ANCOVA — No adjustments made for multiple comparisons; LS mean difference = 0.85, 90% CI 2-sided [-0.75 to 2.45], Standard Error of Mean 0.97
Statistical Analysis 3: Comparison: Placebo vs PF-04447943; Change at Week 9: LS mean difference and p-value were based on ANCOVA on change from baseline with treatment, baseline value, scheduled visit and visit by treatment interaction as covariates, and participant effect as random effect; Test type: Superiority; p = 0.8350, ANCOVA — No adjustments made for multiple comparisons; LS mean difference = 0.96, 90% CI 2-sided [-0.66 to 2.57], Standard Error of Mean 0.98
Statistical Analysis 4: Comparison: Placebo vs PF-04447943; Change at Week 12: LS mean difference and p-value were based on ANCOVA on change from baseline with treatment, baseline value, scheduled visit and visit by treatment interaction as covariates, and participant effect as random effect; Test type: Superiority; p = 0.4377, ANCOVA — No adjustments made for multiple comparisons; LS mean difference = -0.16, 90% CI 2-sided [-1.78 to 1.48], Standard Error of Mean 0.99

7. Other Pre Specified Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Criteria for laboratory test abnormality: a) Hematology: white blood cells (WBC) <0.6*lower limit of normal (LLN)/>1.5*upper limit of normal (ULN), hemoglobin, hematocrit, red blood cells (RBC), lymphocytes <0.8*LLN, total neutrophils <0.8*LLN/ >1.2*ULN, basophils, eosinophils, monocytes >1.2*ULN; b) Liver Function: total bilirubin >1.5*ULN, aspartate aminotransferase (AT), alanine AT[>0.3*ULN, total protein, albumin <0.8*LLN/ >1.2*ULN; c) Renal Function: creatinine >1.3*ULN, uric acid >1.2*ULN; d) Electrolytes: sodium <0.95*LLN/ >1.05*ULN, potassium, chloride, bicarbonate <0.9*LLN/ >1.1*ULN; e) Clinical Chemistry: glucose <0.6*LLN/ >1.5*ULN, glycosylated hemoglobin >1.3*ULN; f) Urinalysis: ketones, protein, blood/hemoglobin, urine glucose >=1, RBC, WBC >=6, hyaline casts >1; g) Hormones: tetraiodothyronine (T4), triiodothyronine (T3) and thyroid stimulating hormone (TSH) <0.8*LLN/1.2*ULN.
Time Frame: Baseline up to Week 12
Population: Safety analysis set included all participants who consumed at least 1 dose of the investigational or control drug. Here, "Overall Number of Participants Analyzed" signifies number of participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-04447943
Number analyzed (Participants) | 99 | 88
Participants | 33 | 28

8. Other Pre Specified Outcome: Number of Participants With Pre-defined Criteria for Electrocardiogram (ECG) Abnormalities
Description: Criteria for ECG (12-lead) abnormalities were as follow: 1) PR interval: greater than and equal to (>=) 300 milliseconds (msec), 2) PR interval: maximum increase from baseline >=25 percent (%) (if baseline PR interval greater than [>] 100 msec) or >=50% (if baseline PR interval less than or equal to [<=] 100 msec); 3) QRS complex: >=200 msec, 4) QRS complex: maximum increase from baseline >=25% or >=50%; 5) QT interval >=500 msec; 6) QT interval corrected using Bazett's formula (QTcB): 450 to less than (<) 480 msec, 7) QTcB: 480 to <500 msec, 8) QTcB: >=500 msec, 10) QTcB: 30 to <60 msec increase from baseline, 11) QTcB: >=60 msec increase from baseline; 9) QT interval corrected using the Fridericia's formula (QTcF): 450 to <480 msec, 10) QTcF: 480 to < 500 msec, 11) QTcF: >=500 msec, 12) QTcF: 30 to <60 msec increase from baseline, 13) QTcF: change>=60 msec increase from baseline.
Time Frame: Baseline up to Week 12
Population: Safety analysis set included all participants who consumed at least 1 dose of the investigational or control drug. Here, "Number Analyzed" signifies those participants who were evaluable for specified rows for each arm, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-04447943
Number analyzed (Participants) | 100 | 91
Participants
  PR interval >=300 msec: number analyzed (Participants) | 99 | 88
  PR interval >=300 msec | 0 | 0
  PR interval: 25% or 50% increase: number analyzed (Participants) | 94 | 83
  PR interval: 25% or 50% increase | 0 | 0
  QRS complex >=200 msec: number analyzed (Participants) | 99 | 91
  QRS complex >=200 msec | 0 | 1
  QRS interval: >=25% or 50% increase: number analyzed (Participants) | 95 | 87
  QRS interval: >=25% or 50% increase | 1 | 1
  QT interval >=500 msec: number analyzed (Participants) | 99 | 91
  QT interval >=500 msec | 2 | 1
  QTcB interval: 450 to < 480 msec: number analyzed (Participants) | 99 | 91
  QTcB interval: 450 to < 480 msec | 19 | 22
  QTcB interval: 480 to < 500 msec: number analyzed (Participants) | 99 | 91
  QTcB interval: 480 to < 500 msec | 4 | 1
  QTcB interval >= 500 msec: number analyzed (Participants) | 99 | 91
  QTcB interval >= 500 msec | 0 | 3
  QTcB interval: 30 to <60 msec increase: number analyzed (Participants) | 95 | 86
  QTcB interval: 30 to <60 msec increase | 11 | 13
  QTcB interval: >=60 msec increase: number analyzed (Participants) | 95 | 86
  QTcB interval: >=60 msec increase | 0 | 1
  QTcF interval: 450 to <480 msec: number analyzed (Participants) | 99 | 91
  QTcF interval: 450 to <480 msec | 9 | 12
  QTcF interval: 480 to <500 msec: number analyzed (Participants) | 99 | 91
  QTcF interval: 480 to <500 msec | 4 | 0
  QTcF Interval >= 500 msec: number analyzed (Participants) | 99 | 91
  QTcF Interval >= 500 msec | 0 | 3
  QTcF interval: 30 to <60 msec increase: number analyzed (Participants) | 95 | 86
  QTcF interval: 30 to <60 msec increase | 6 | 10
  QTcF interval: >=60 msec increase: number analyzed (Participants) | 95 | 86
  QTcF interval: >=60 msec increase | 2 | 1

9. Other Pre Specified Outcome: Number of Participants With Abnormal Physical Examinations and Neurological Examinations
Description: The complete physical and neurological examination included examination of abdomen, ears, extremities, eyes, general, head, heart, lungs, lymph nodes, mouth, musculoskeletal, neck, nose, ocular fundi, pulse, skin, throat, thyroid, and others. Abnormality was judged by investigator.
Time Frame: Screening (28 days before Baseline), Week 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-04447943
Number analyzed (Participants) | 100 | 91
Participants
  Abdomen: Screening: number analyzed (Participants) | 100 | 89
  Abdomen: Screening | 9 | 9
  Abdomen: Week 12: number analyzed (Participants) | 96 | 86
  Abdomen: Week 12 | 5 | 6
  Ears: Screening: number analyzed (Participants) | 99 | 91
  Ears: Screening | 6 | 9
  Ears: Week 12: number analyzed (Participants) | 95 | 86
  Ears: Week 12 | 3 | 9
  Extremities: Screening: number analyzed (Participants) | 98 | 86
  Extremities: Screening | 15 | 15
  Extremities: Week 12: number analyzed (Participants) | 95 | 86
  Extremities: Week 12 | 10 | 11
  Eyes: Screening | 26 | 26
  Eyes: Week 12: number analyzed (Participants) | 96 | 86
  Eyes: Week 12 | 24 | 22
  General: Screening | 1 | 2
  General: Week 12: number analyzed (Participants) | 96 | 86
  General: Week 12 | 2 | 2
  Head: Screening: number analyzed (Participants) | 99 | 91
  Head: Screening | 1 | 1
  Head: Week 12: number analyzed (Participants) | 95 | 86
  Head: Week 12 | 1 | 1
  Heart: Screening: number analyzed (Participants) | 100 | 90
  Heart: Screening | 3 | 8
  Heart: Week 12: number analyzed (Participants) | 96 | 86
  Heart: Week 12 | 3 | 5
  Lungs: Screening | 3 | 0
  Lungs: Week 12: number analyzed (Participants) | 96 | 86
  Lungs: Week 12 | 3 | 0
  Lymph nodes: Screening: number analyzed (Participants) | 92 | 84
  Lymph nodes: Screening | 0 | 0
  Lymph nodes: Week 12: number analyzed (Participants) | 96 | 85
  Lymph nodes: Week 12 | 0 | 1
  Mouth: Screening: number analyzed (Participants) | 100 | 90
  Mouth: Screening | 11 | 3
  Mouth: Week 12: number analyzed (Participants) | 96 | 86
  Mouth: Week 12 | 9 | 3
  Musculoskeletal: Screening: number analyzed (Participants) | 99 | 91
  Musculoskeletal: Screening | 11 | 13
  Musculoskeletal: Week 12: number analyzed (Participants) | 96 | 86
  Musculoskeletal: Week 12 | 7 | 12
  Neck: Screening | 1 | 2
  Neck: Week 12: number analyzed (Participants) | 96 | 86
  Neck: Week 12 | 0 | 0
  Nose: Screening: number analyzed (Participants) | 98 | 91
  Nose: Screening | 0 | 2
  Nose: Week 12: number analyzed (Participants) | 95 | 86
  Nose: Week 12 | 0 | 1
  Ocular fundi: Screening: number analyzed (Participants) | 85 | 73
  Ocular fundi: Screening | 1 | 2
  Ocular fundi: Week 12: number analyzed (Participants) | 85 | 75
  Ocular fundi: Week 12 | 1 | 0
  Pulses: Screening: number analyzed (Participants) | 97 | 90
  Pulses: Screening | 2 | 3
  Pulses: Week 12: number analyzed (Participants) | 96 | 86
  Pulses: Week 12 | 0 | 0
  Skin: Screening | 30 | 23
  Skin: Week 12: number analyzed (Participants) | 95 | 86
  Skin: Week 12 | 25 | 21
  Throat: Screening: number analyzed (Participants) | 99 | 91
  Throat: Screening | 0 | 0
  Throat: Week 12: number analyzed (Participants) | 96 | 86
  Throat: Week 12 | 0 | 0
  Thyroid: Screening: number analyzed (Participants) | 100 | 88
  Thyroid: Screening | 0 | 3
  Thyroid: Week 12: number analyzed (Participants) | 96 | 85
  Thyroid: Week 12 | 0 | 3
  Other: Screening: number analyzed (Participants) | 25 | 24
  Other: Screening | 2 | 1
  Other: Week 12: number analyzed (Participants) | 13 | 17
  Other: Week 12 | 0 | 3

10. Other Pre Specified Outcome: Number of Participants With Categorical Scores on the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS assessed whether participant experienced the following: suicidal behavior which includes suicide attempt, interrupted attempt, aborted attempt, and preparatory acts towards imminent suicidal behavior (response of "Yes" on "preparatory acts or behavior"); suicidal ideation (response of "Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent); self-injurious behavior (SIB), intent unknown (response of "Yes" on "Has subject engaged in Non-suicidal Self-Injurious Behavior?").
Time Frame: Screening, Baseline, Post-baseline (Week 1 up to 12)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-04447943
Number analyzed (Participants) | 100 | 91
Participants
  Suicidal behavior: Screening | 0 | 0
  Suicide attempt: Screening | 0 | 0
  Interrupted attempt: Screening | 0 | 0
  Aborted attempt: Screening | 0 | 0
  Imminent suicidal behavior: Screening | 0 | 0
  Suicidal ideation: Screening | 5 | 6
  Non-suicidal SIB: Screening | 0 | 0
  Suicidal behavior: Baseline | 0 | 0
  Suicide attempt: Baseline | 0 | 0
  Interrupted Attempt: Baseline | 0 | 0
  Aborted attempt: Baseline | 0 | 0
  Imminent suicidal behavior: Baseline | 0 | 0
  Suicidal ideation: Baseline | 4 | 5
  Non-Suicidal SIB: Baseline | 0 | 0
  Suicidal behavior: Post baseline: number analyzed (Participants) | 100 | 89
  Suicidal behavior: Post baseline | 0 | 0
  Suicide attempt: Post baseline: number analyzed (Participants) | 100 | 89
  Suicide attempt: Post baseline | 0 | 0
  Interrupted attempt: Post baseline: number analyzed (Participants) | 100 | 89
  Interrupted attempt: Post baseline | 0 | 0
  Aborted attempt: Post baseline: number analyzed (Participants) | 100 | 89
  Aborted attempt: Post baseline | 0 | 0
  Imminent suicidal behavior:Post baseline: number analyzed (Participants) | 100 | 89
  Imminent suicidal behavior:Post baseline | 0 | 0
  Suicidal ideation: Post baseline: number analyzed (Participants) | 100 | 89
  Suicidal ideation: Post baseline | 6 | 6
  Non-suicidal SIB: Post baseline: number analyzed (Participants) | 100 | 89
  Non-suicidal SIB: Post baseline | 0 | 1

11. Other Pre Specified Outcome: PF-04447943 Plasma Concentration
Time Frame: Pre-dose on Week 1; 0 to 3 hours following cognitive testing at Week 3, 6, 9, 12
Population: FAS included all the participants who consumed at least 1 dose of randomized study medication. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this measure and "Number Analyzed" signifies those participants who were evaluable for this measure at the specified time points.
Measure: Median (Full Range); unit: nanogram per milliliter
Arm/Group | Placebo | PF-04447943
Number analyzed (Participants) | 90 | 80
nanogram per milliliter
  Week 1: number analyzed (Participants) | 1 | 79
  Week 1 | NA [NA to NA] — Data was not estimable as none of the participants had concentration above than lower limit of quantification. | 71.60 [0.000 to 407]
  Week 3: number analyzed (Participants) | 1 | 80
  Week 3 | NA [NA to NA] — Data was not estimable as none of the participants had concentration above than lower limit of quantification. | 241.0 [0.000 to 561]
  Week 6: number analyzed (Participants) | 1 | 79
  Week 6 | NA [NA to NA] — Data was not estimable as none of the participants had concentration above than lower limit of quantification. | 225.0 [0.000 to 693]
  Week 9 | 0.0000 [0.0 to 40.6] | 239.5 [0.000 to 738]
  Week 12: number analyzed (Participants) | 1 | 80
  Week 12 | NA [NA to NA] — Data was not estimable as none of the participants had concentration above than lower limit of quantification. | 250.5 [0.000 to 598]

12. Other Pre Specified Outcome: Number of Participants With Pre-defined Criteria of Vital Signs Abnormalities
Description: Pre-defined criteria vital signs abnormalities included maximum increase or decrease of greater than or equal to (>=) 30 millimeters of mercury (mmHg) from baseline for supine systolic blood pressure (SBP); maximum increase or decrease of >=20 mmHg from baseline for supine diastolic BP (DBP); maximum increase or decrease of >=30 mmHg from baseline for standing SBP; maximum increase or decrease of >=20 mmHg from baseline for standing DBP. Orthostatic hypotension was defined as a drop of more than 10 mmHg in diastolic BP or a drop of more than 20 mmHg in systolic BP within 3 minutes of standing from the supine position.
Time Frame: Baseline up to Week 12 for change in supine or standing blood pressure; Week 1, 3, 6, 9, 12 for orthostatic hypotension
Population: Safety analysis set included all participants who consumed at least 1 dose of the investigational or control drug. "Number Analyzed" signifies those participants who were evaluable for the specified rows for each arm, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-04447943
Number analyzed (Participants) | 100 | 91
Participants
  Increase in supine SBP (>=30 mmHg): number analyzed (Participants) | 100 | 89
  Increase in supine SBP (>=30 mmHg) | 9 | 4
  Decrease in supine SBP (>=30 mmHg): number analyzed (Participants) | 100 | 89
  Decrease in supine SBP (>=30 mmHg) | 5 | 8
  Increase in standing SBP (>=30 mmHg): number analyzed (Participants) | 100 | 88
  Increase in standing SBP (>=30 mmHg) | 6 | 7
  Decrease in Standing SBP (>=30 mmHg): number analyzed (Participants) | 100 | 88
  Decrease in Standing SBP (>=30 mmHg) | 11 | 9
  Increase in supine DBP (>=20 mmHg): number analyzed (Participants) | 100 | 89
  Increase in supine DBP (>=20 mmHg) | 3 | 2
  Decrease in Supine DBP (>=20 mmHg) (: number analyzed (Participants) | 100 | 89
  Decrease in Supine DBP (>=20 mmHg) ( | 9 | 8
  Increase in standing DBP(>=20 mmHg): number analyzed (Participants) | 100 | 88
  Increase in standing DBP(>=20 mmHg) | 4 | 3
  Decrease in Standing DBP(>=20 mmHg): number analyzed (Participants) | 100 | 88
  Decrease in Standing DBP(>=20 mmHg) | 4 | 6
  Orthostatic Hypotension: Week 1 | 5 | 3
  Orthostatic Hypotension: Week 3 | 3 | 3
  Orthostatic Hypotension: Week 6 | 4 | 2
  Orthostatic Hypotension: Week 9 | 2 | 4
  Orthostatic Hypotension: Week 12 | 5 | 4

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | PF-04447943
Serious Adverse Events (participants affected / at risk) | 4/100 | 3/91
Other Adverse Events (participants affected / at risk) | 56/100 | 57/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=100) | PF-04447943 (N=91)
Cardiac arrest (Cardiac disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Chronic hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=100) | PF-04447943 (N=91)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Bundle branch block right (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 4 | 2
Conjunctivitis (Eye disorders) | 1 | 0
Eyelid irritation (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 5
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 2 | 0
Chest pain (General disorders) | 0 | 2
Fatigue (General disorders) | 1 | 1
Irritability (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 2 | 1
Seasonal allergy (Immune system disorders) | 1 | 0
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0
Bacteriuria (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 2 | 3
Cellulitis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 3
Labyrinthitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 5 | 4
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 2
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1
Stab wound (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 2 | 3
Blood pressure decreased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Blood sodium increased (Investigations) | 0 | 1
Carotid bruit (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Headache (Nervous system disorders) | 7 | 7
Neuralgia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Poor quality sleep (Nervous system disorders) | 0 | 1
Sedation (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 2 | 3
Tension headache (Nervous system disorders) | 2 | 0
Abnormal behaviour (Psychiatric disorders) | 1 | 1
Aggression (Psychiatric disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Depressed mood (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Eating disorder (Psychiatric disorders) | 0 | 1
Initial insomnia (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 4
Nightmare (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Glycosuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Pyuria (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 1
Right Knee Sore (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.